CLINICAL TRIAL: NCT01276795
Title: Whey Protein-based Enteral Nutrition Support to Improve Protein Economy in Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other)
Responsible Party: Dr. Francesco Carli, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-053-SDR
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2010-07

CONDITIONS: Protein Metabolism; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucose and whey protein (Experimental): Patients who are randomly allocated to this group will receive a drink made of anhydrous beet dextrose and pressurized whey protein in water (200 g/L + 100g/L). Patients will sip the drink for 4 hours of the 6 hour study.
  Interventions: Dietary Supplement: Oral Nutrition Support
- Glucose only (Active Comparator): The patients who are randomly allocated to this arm will receive a drink composed of anhydrous beet dextrose in water (200g/L). They will sip the drink for 4 hours of the 6 hour study.
  Interventions: Dietary Supplement: Oral Nutrition Support

INTERVENTIONS:
Dietary Supplement: Oral Nutrition Support — The patients will sip the oral nutrition support (in the form of a drink) over the course of 4 hours within each 6 hour study. Each patient will be studied once before surgery and once after surgery.

SUMMARY:
A prospective, randomized and controlled study is proposed to establish whether an enteral nutrition support regimen based on pressurized whey protein and glucose improves the postoperative utilization of amino acid substrates compared to a drink based on glucose alone. The kinetics of protein metabolism (protein breakdown, protein synthesis and amino acid oxidation) will be investigated using stable isotope methodology before and after surgery in patients undergoing colon resection. Stable isotope infusions will be conducted one week before surgery and on the second postoperative day for two hours in the fasted state and for four hours while sipping the enteral nutrition support regimen. Patients will consume one of two enteral nutrition support regimens consisting of a drink containing either pressurized whey protein and glucose or glucose alone. It is hypothesized that an enteral nutrition support regimen based on pressurized whey protein and glucose promotes positive protein balance through increased protein synthesis or reduced protein breakdown compared to glucose alone.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* ASA class I to III
* colorectal surgery for non-metastatic disease (including right, transverse, left, sigmoid, subtotal, total and hemicolectomy and low anterior resection)
* body mass index >17 and <30 kg.m-2
* stable weight over the preceding three months (<10 % body weight loss)
* serum albumin >35 g/L

Exclusion Criteria:

* severe cardiac, renal or hepatic failure
* diabetes
* hyper and hypothyroidism
* active inflammatory bowel or diverticular disease
* musculoskeletal or neuromuscular disease
* anemia (hematocrit <30)
* albumin < 25 g/l
* pregnancy
* use of steroids.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Protein balance | Assessed for 6 hours one time before surgery and once again on the second post-op day
  Protein balance is assessed using the stable isotope tracer C-13 leucine. Protein breakdown, protein synthesis and amino acid oxidation are measured through blood and expired air samples.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD PhD, Principal Investigator — McGill University
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada